CLINICAL TRIAL: NCT01514006
Title: Postoperative Anemia and Functional Outcomes After Fast-track Primary Hip Arthroplasty - a Prospective Observational Study
Brief Title: Postoperative Anemia and Functional Outcomes After Fast-track Primary Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other); Vejle Hospital (Other)
Responsible Party: Principal Investigator, Oeivind Jans, MD., Research Fellow, Rigshospitalet, Denmark
Other Study IDs: H-4-2011-117
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Arthroplasty, Hip Replacement; Anemia
Keywords: Primary hip arthroplasty; postoperative anemia; functional outcomes
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Cohort: Patients, aged 65 or above, undergoing elective primary unilateral hip arthroplasty in a fast-track setting.

SUMMARY:
The purpose of this study is to evaluate the possible association between postoperative anaemia and functional outcomes the first 2 weeks after primary hip arthroplasty.

The investigators hypothesise that patients with a higher degree of postoperative anaemia have impaired postoperative rehabilitation as measured by standardized functional outcome tests.

DETAILED DESCRIPTION:
Postoperative anemia may impair postoperative rehabilitation due to anemia related symptoms such as fatigue or dizziness. Although, the impact of postoperative anemia on postoperative rehabilitation and function has previously been examined the results are conflicting.

Patients undergoing fast-track hip arthroplasty (THA) are mobilized early and participate in physiotherapy during the admission but are discharged early (2-3) days postoperative. However, the ability to rehabilitate early after discharge has not been evaluated in relation to postoperative anemia.

The purpose of this observational study is to evaluate the possible association between postoperative anaemia and functional outcomes the first 2 weeks after primary hip arthroplasty.

The investigators hypothesise that patients with a higher degree of postoperative anaemia have impaired postoperative rehabilitation as measured by standardized functional outcome tests. Hb concentrations and functional outcome measurements will be performed preoperatively, at the day of hospital discharge and during a postoperative visit 12-16 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary unilateral THA
* Age 65 or older

Exclusion Criteria:

* Not able to give consent
* Not able to walk prior to surgery
* Chronic need for RBC transfusion

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients aged 65 or above undergoing primary hip arhtroplasty
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
6 Minute walking test (6MWT) | 2 weeks after surgery
  6MWT is a standardized functional test which determines the walking distance covered during a timed period of 6 minutes.

SECONDARY OUTCOMES:
FACT-Anemia Scale | 2 weeks after surgery
  FACT-Anemia scale is a validated questionare based score addressing anaemia related symptoms.
Timed up and go test (TUG) | 2 weeks after surgery
At home activity by ActivPal | 1 week after surgery
  Activity measures using accelerometer based activity monitor

CONTACTS AND LOCATIONS:
Overall Officials: Oeivind Jans, MD., Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Gentofte Hospital, Department of orthopedic surgery, Gentofte Municipality
  - Vejle Sygehus, Department of orthopedic surgery, Vejle